CLINICAL TRIAL: NCT06901869
Title: ActivPARK - Physical Activity in Persons With Parkinson's Disease- Pilot Study
Brief Title: Physical Activity in Persons With Parkinson's Disease
Acronym: ActivPARK
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Lund University (Other); Göteborg University (Other); Umeå University (Other); Region Stockholm (Other Government); Vastra Gotaland Region (Other Government); Region Skane (Other); Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Erika Franzén, Professor, Karolinska Institutet
Other Study IDs: 2024-07526-01; 2024-06332 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2025-03-17; First posted 2025-03-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Physical Inactivity
MeSH Terms: conditions — Parkinson Disease; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Parkinson's disease: No intervention

SUMMARY:
Parkinson's disease (PD) is a leading neurodegenerative health condition in Sweden and a public health concern. Although no cure exists, functional independence and participation in society remain top priorities, and can be achieved through targeted physical activity (PA) interventions. To date, few longitudinal cohort studies have been conducted, using PA as main outcome in therapy research, partly due to the complex nature of predicting and controlling this phenomenon. To help address this knowledge gap, the overall purpose of the future long-term (ActivPARK) study is to enhance knowledge of the evolution of PA behavior, and how it is influenced beyond the disease characteristics using a broad explanatory model, in persons with PD from a diversity of settings in Sweden with the aim of prescribing tailored and personalized interventions to enhance functioning, health, and wellbeing throughout the disease progression and recommend potential health care pathway modifications.

The investigators have just established an expert group, comprising researchers, healthcare professionals, and PD organisations (including persons with PD) and reached consensus on essential priority clinical therapy research questions on PA and methodological considerations. The next phase entails performing a multicentre feasibility/pilot study, further developing and refining the assessment battery and research questions linked to the improved explanatory model for PA and methodology, to inform the definite larger clinical cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease
* Mild to severe disease severity ( Hoehn & Yahr 1-4).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's disease with mild to severe severity (Hoehn & Yahr 1-4) of all ages
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the assessment battery - length of the clinical examination and questionnaires | Baseline
  The pilot/feasibility study aims to evaluate feasibility of the assessment battery measured the time it takes to complete the examination and questionnaires.
Feasibility of the assessment battery - perception of the clinical examination | Baseline
  Feasibility of the assessment battery will also be evaluated through semi-structured questions regarding fatique, concentration, pain/discomfort to the participants after the clinical examination.
Feasibility of the assessment battery -Compliance to questionnaires sent via REDCap | Baselline
  Compliance will be measured with percentages of completed questionnaires in REDCap.
Feasibility of the assessment battery - Suitability of the primary outcome | Baseline
  Suitability of the accelerometers in the home environment as the primary outcome for the targeted patient group will be assessed by the percentage of participants that are able to wear the accelerometer for at least 4 days days and render valid data.
Physical activity levels | Baseline
  The ActiGraph accelerometer (GT3X+, ActiGraph, Pensacola, FL, US) will be used to measure absolute and relative time spent in sedentary behavior, low intensity physical activity (LIPA) and moderate to vigorous intensity physical activity (MVPA), by total time in bouts.

SECONDARY OUTCOMES:
Physical activity - self rated | Baseline
  Frändin Grimby scale, ranging from 1 to 6, higher score=better.
Disease severity, Parkinson symptoms | Baseline
  Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS- UPDRS) parts 1 to 4.
  Higher scores = worse/more symptoms
Gait | Baseline
  Gait speed in m/s measured with the 10 meter walking test or through gait analysis.
Balance performance | Baseline
  Assessed with the Mini-BESTest. Mini-Balance Evaluation Systems Test a rating scale for dynamic balance incorporating 14 different balance and gait items that were assessed by a physical therapist on a scale from 0-2. Maximum points 28. 0-28 points with higher scores indicating better balance control
Anxiety and depression | Baseline
  Assessed with Hospital Anxiety and Depression Scale (HADS), 0-24 on the depression and anxiety part respectively. Lower score=better
Cognitive performance | Baseline and 3 year follow-up
  Assessed with the Montreal Cognitive Assessment (MoCA), 0-25, higher score = better
Self assessed cognitive function | Baseline
  Assessed with Executive function questionnaire (DEX), 20 items scored 1 to 4, max 80, more scores= worse.
Non-Motor Symptoms | Baseline
  Non-Motor Symptoms Questionnaire (NMSQ), 30 questions with yes/no answer. More yes answers = more non-motor symptoms
Walking ability- self assessed | Baseline
  WALK-12G questionnaire, 0 and 42 points, with higher scores reflecting greater perceived walking difficulties (higher=worse)
Freezing of gait - self-assessed | Baseline
  Freezing of gait questionnaire (FOGQsa), 6 questions/items, scored 1 to 5 (higher=worse)
Balance confidence | Baseline
  Activities specific balance confidence (ABC scale), 16 items which is scored 1 to 10 and then divided by 16. 0-100%, higher % = better
Motivation | Baseline
  Behavioural Regulation in Exercise Questionnaire (BREQ 4), 28 items score 1 to 7 and divided into subcomponents: Amotivation, External regulation, Introjected avoidance, Introjected approach, Identified regulation, Integrated regulation, Intrinsic regulation
Fatigue | Baseline
  Parkinson's Fatigue Scale (PFS-16), 16 items scored 1 to 5 from strongly disagree to strongly agree . more points/score= worse.
Disability | Baseline
  World health organization (WHO) disability assessment schedule (Whodas 2.0), 12 self-assessed questions (12 to 60) more points=worse
Self-efficacy | Baseline
  Self-efficacy of exercise/PA (ESES), 10 questions, scored 1-4. higher=better
Sleep | Baseline
  Scales for Outcomes in Parkinson's disease - Sleep (SCOPA-SLEEP), 4 parts, A-2 questions, B-5 questions , C-1 question and D- 6 questions. Higher= worse
Self rated pain | Baseline
  Assessed with visual analog scale, VAS from 0 to 100
Health related quality of life | Baseline
  Parkinson's Disease Questionnaire (PDQ39). The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communications and bodily discomfort). The sum score is as a percentage score ranging between 0 and 100. Higher is better
Wellbeing | Baseline
  The WHO- Five Well-Being Index (WHO-5), 5 questions ranging from 0 to 5, 0-25, higher=better
Nutrition | Baseline
  Mini Nutritional Assessment, max 14. higher = better

OTHER OUTCOMES:
Working och long-term memory | Baseline
  Rey-Auditory Verbal Learning Test (RAVLT), higher= better
Parkinson related pain | Baseline
  Assessed with the Kings Parkinsons Pain Scale (KPPS), max 168, higher= more pain

CONTACTS AND LOCATIONS:
Overall Officials: Erika Franzén, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient, provided that the recipient has an approved ethics application.
Supporting Information: SAP
Time Frame: The investigators plan to share this when applicable on OSF or similar
Access Criteria: The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT06901869/Prot_SAP_000.pdf